CLINICAL TRIAL: NCT00486044
Title: Effect of Statins on Pathobiology of Alzheimer's Disease
Brief Title: Evaluating Simvastatin's Potential Role in Therapy
Acronym: ESPRIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Paul Beeson Faculty Scholars Program (Other); The John A. Hartford Foundation (Other); The Atlantic Philanthropies (Other); Starr Foundation (Other); American Federation for Aging Research (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IA0116; 1K23AG026752-01 (NIH)
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer Disease
Keywords: amyloid protein; apolipoprotein; cerebrospinal fluid; cerebrovascular circulation; inflammation; magnetic resonance imaging; prevention & control
MeSH Terms: conditions — Alzheimer Disease; Amyloidosis; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simvastatin (Experimental): simvastatin 40 mg nightly for 1 month then 80 mg nightly for 8 months
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Matching placebo tablet nightly for 9 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg tablet each night for one month, then 80 mg for 8 months
  Other Names: Zocor
  Arms: simvastatin
Drug: Placebo — Matching tablet each night for 9 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to see how simvastatin, a cholesterol-lowering drug, affects processes related to the development of Alzheimer's disease, including: 1) levels of a substance called beta-amyloid-42 found in the spinal fluid surrounding the brain, 2) blood flow in the brain, 3) inflammation in the brain, and 4) cognitive function.

DETAILED DESCRIPTION:
Some studies suggest that statin medications, which are a group of cholesterol-lowering medicines, may help prevent Alzheimer's disease. However, this has not been proven in humans. The purpose of this study is to see how simvastatin affects a substance in the spinal fluid around the brain called beta-amyloid-42 which is thought to contribute to Alzheimer's disease. This study also evaluates whether simvastatin improves regional brain blood flow (on magnetic resonance imaging [MRI]), reduces inflammation, and improves cognitive function.

The ESPRIT study was a 9-month randomized, controlled clinical trial that randomized 100 middle-aged adults with a parental history of Alzheimer's disease. Participants were randomized to simvastatin 40 mg for one month then 80 mg daily or matching placebo tablets. Fifty of the ESPRIT subjects participated in the MRI sub-study.

Participants had the following data collected: fasting blood tests (baseline and months 3 and 9), medical history and medication questionnaires (each visit), study medication side effect review (all visits), lumbar puncture procedure (baseline and month 9), memory testing (baseline and months 3 and 9), and MRI (baseline and month 9 in 50 sub-study participants).

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 69
* Parent with Alzheimer's disease

Exclusion Criteria:

* Current use of cholesterol-lowering medication
* Active liver disease
* History of adverse reaction to statins
* Contraindication to lumbar puncture
* Elevated lab values (creatine kinase and creatinine)
* Use of medications known to interact with statins
* History of dementia
* Currently pregnant or planning to become pregnant
* Use of large quantities of grapefruit juice (more than 1 quart per day)
* Current involvement in another investigational drug study
* Contraindications to MRI (for MRI sub-study)
* Ethical contraindication to placebo (persons with high vascular risk)

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M. Carlsson, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Fassbender K, Simons M, Bergmann C, Stroick M, Lutjohann D, Keller P, Runz H, Kuhl S, Bertsch T, von Bergmann K, Hennerici M, Beyreuther K, Hartmann T. Simvastatin strongly reduces levels of Alzheimer's disease beta -amyloid peptides Abeta 42 and Abeta 40 in vitro and in vivo. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5856-61. doi: 10.1073/pnas.081620098. Epub 2001 Apr 10. PMID 11296263
- [Background] Wolozin B. A fluid connection: cholesterol and Abeta. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5371-3. doi: 10.1073/pnas.101123198. No abstract available. PMID 11344276
- [Background] Johnson NA, Jahng GH, Weiner MW, Miller BL, Chui HC, Jagust WJ, Gorno-Tempini ML, Schuff N. Pattern of cerebral hypoperfusion in Alzheimer disease and mild cognitive impairment measured with arterial spin-labeling MR imaging: initial experience. Radiology. 2005 Mar;234(3):851-9. doi: 10.1148/radiol.2343040197. PMID 15734937
- See also: Wisconsin Alzheimer's Disease Research Center — http://adrc.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Middle-aged adults with parental history of Alzheimer's disease were recruited for this single-site trial (Madison, Wisconsin) from the Wisconsin Registry for Alzheimer's Prevention (WRAP) or the community through newsletters, websites, educational talks, health fairs, local clinics, and newspaper and magazine advertisements.
Pre-assignment Details: 103 participants enrolled in the trial and 100 were randomized to treatment (1 no longer met inclusion criteria, 2 declined participation).
Groups:
- Simvastatin: Simvastatin 40 mg tablet nightly for 1 month then 80 mg tablet nightly for 8 months
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 51 (50 received assigned intervention (1 withdrew during baseline) 27 in MRI sub-study) | 49 (23 in MRI sub-study)
Completed | 49 (27 completed MRI sub-study) | 46 (21 completed MRI sub-study)
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 42 | 91
  >=65 years | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (7.4) | 52.4 (8.5) | 52.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100
Education [Mean (Standard Deviation); unit: years] | 16.1 (2.) | 16.3 (3.2) | 16.2 (2.9)
Cognitive Function [Mean (Standard Deviation); unit: points] — Measured by Mini Mental State Exam (MMSE), a cognitive battery scored on a 0-30 point range where >24 points indiacte better outcomes; <24 points indicates cognitive dysfunction.
  points | 29.5 (0.8) | 29.6 (0.6) | 29.5 (0.7)
Apolipoprotein E4 carrier [Number; unit: participants] — Apolipoprotein E4 (APOE4) carrier status was determined by genotyping whole blood from subjects.
  participants | 21 | 17 | 38
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] — Measured by nuclear magnetic resonance (NMR) spectroscopy
  mg/dL | 192.8 (36.4) | 187.6 (27.7) | 190.3 (32.4)
High-sensitivity c-reactive protein [Mean (Standard Deviation); unit: mg/L] | 2.59 (3.71) | 2.03 (2.21) | 2.32 (3.06)
Cerebrospinal fluid beta-amyloid-42 [Mean (Standard Deviation); unit: ng/L] — Cerebrospinal fluid beta amyloid 42 was measured by XMAP.
  ng/L | 345.6 (77.1) | 331.0 (83.7) | 338.7 (80.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebrospinal Fluid (CSF) Beta-amyloid-42
Time Frame: baseline and 9 months
Population: 1 participant declined follow up CSF collection in simvastatin arm; CSF could not be accessed at month 9 in 1 participant in placebo arm
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 48 | 45
ng/L | -5.2 (44.1) | -3.1 (38.2)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = 0.966, Kruskal-Wallis

2. Secondary Outcome: Changes in Regional Cerebral Blood Flow on MRI
Description: Mean changes noted in posterior cingulate cortex
Time Frame: baseline and 9 months
Population: Number of participants analyzed represent participants in MRI substudy with readable MRI scans at both baseline and 9 months; 24 and 17 readable MRI scans in simvastatin and placebo arms, respectively. Unusable MRI scans resulted from poor quality images due to technical problems.
Measure: Mean (Standard Deviation); unit: mL/100 g/min
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 24 | 17
mL/100 g/min | 4.09 (6.69) | -5.08 (8.28)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA

3. Secondary Outcome: Change in Inflammatory Markers
Description: Change noted in serum high-sensitivity c-reactive protein
Time Frame: baseline and 9 months
Population: 2 participants in the simvastatin arm and 3 participants in the placebo arm had incomplete hs-CRP results
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 47 | 43
mg/L | -1.16 (3.55) | -0.31 (1.83)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = 0.113, Kruskal-Wallis

4. Secondary Outcome: Changes in Cognitive Performance
Description: Change in Hopkins Verbal Learning Test Delayed Recall
  The Hopkins Verbal Learning Test Delayed Recall score is the raw number of words recalled at Trial 4, adjusted for years of education and age. This is a 12-item word list test.
Time Frame: Baseline and 9 months
Population: 1 participant in simvastatin arm with missing data
Measure: Mean (Standard Deviation); unit: adjusted words recalled
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 48 | 46
adjusted words recalled | 0.40 (1.38) | 0.26 (1.54)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = 0.210, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 4/51 | 1/49
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=51) | Placebo (N=49)
Elevated creatine kinase (CK) (> 2 times upper limit of normal) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Elevated liver transaminases (>2 times upper limit of normal) (Hepatobiliary disorders) | 2 (2) | 0 (0)
Anxiety/depression (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No